CLINICAL TRIAL: NCT05604872
Title: Association Between Preoperative Ocular Residual Astigmatism(ORA) and Residual Refractive Astigmatism After SMILE Refractive Surgery
Brief Title: Association Between ORA and Residual Refractive Astigmatism After SMILE
Status: Completed | Type: Observational
Sponsor: Taipei Nobel Eye Clinic (Other)
Responsible Party: Principal Investigator, Chao-Kai Chang, Dean, Taipei Nobel Eye Clinic
Other Study IDs: 003
Record Dates: First submitted 2022-10-31; First posted 2022-11-03 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-10

CONDITIONS: Refractive Errors; Astigmatism
MeSH Terms: conditions — Refractive Errors; Astigmatism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Small Incision Lenticule Extraction — A 500 kHzVisumax (Carl Zeiss Meditec AG) femtosecond laser was used with cap thickness ranging from 100 to 130μm, cap diameter from 7.3 to 7.9 mm. The lenticule was dissected with a blunt spatula through a 30 to 60-degree incision at the 10 o'clock position and removed using forceps afterward. Treatment targets of both eyes were set to emmetropia, the refraction corrections were based on manifest refractions

SUMMARY:
The aim of our study is to analysis and compare the relationship between ORA and postoperative astigmatism in low astigmatism (less than 1D) and moderate to high (1D to 3D) astigmatism patients after SMILE (Small Incision Lenticule Extraction) refractive surgery.

ELIGIBILITY:
Inclusion Criteria:

* Corrected distance visual acuity of both eyes reaches 0.1 logarithm of the minimum angle of resolution (logMAR)
* Stable refractive errors of myopia and astigmatism who received SMILE refractive surgery of both eyes

Exclusion Criteria:

* Cataract
* Corneal opacities or irregularities
* Dry eye (Schirmer's test I ≤ 5mm)
* Amblyopia
* Coexisting ocular pathologies
* Glaucoma
* Non-dilating pupil
* History of intraocular surgery, laser therapy, or retinopathy
* Optic nerve or macular diseases
* Estimated postoperative cornea residual stromal thickness less than 250 μm
* Pregnancy or under lactation
* Uncontrolled diabetic mellitus or systemic immune disease _Refusal or unable to maintain follow-up

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: This study was conducted by retrospective chart review in Taipei Nobel Eye Clinic from 2020 to 2022.
Sampling Method: Non-Probability Sample
Enrollment: 530 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Corrected distance visual acuity | 3 months after surgery
  in LogMAR unit
Manifest refraction | 3 months after surgery
  in Diopter

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Nobel Eye Clinic, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gyldenkerne A, Hjortdal J, Ivarsen A. Astigmatism prediction in small-incision lenticule extraction. J Cataract Refract Surg. 2020 Apr;46(4):524-533. doi: 10.1097/j.jcrs.0000000000000083. PMID 32271519
- [Result] Jun I, Kang DSY, Arba-Mosquera S, Reinstein DZ, Archer TJ, Jean SK, Kim EK, Seo KY, Lee HK, Kim TI. Comparison of clinical outcomes between vector planning and manifest refraction planning in SMILE for myopic astigmatism. J Cataract Refract Surg. 2020 Aug;46(8):1149-1158. doi: 10.1097/j.jcrs.0000000000000100. PMID 32347695
- [Derived] Chao CC, Lin MY, Chang CK. The Association Between Ocular Residual Astigmatism and the Efficacy of Astigmatism Correction Via Small Incision Lenticule Extraction (SMILE). Ophthalmol Ther. 2023 Oct;12(5):2631-2640. doi: 10.1007/s40123-023-00766-1. Epub 2023 Jul 20. PMID 37470969